CLINICAL TRIAL: NCT03518970
Title: Nursing Intervention to Manage Uncertainty in Illness in Palliative Care: Feasibility and Acceptability Study in Family Caregivers
Brief Title: Uncertainty in Illness in Palliative Care: an Intervention for Family Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AVAL-O35-17
Record Dates: First submitted 2018-04-15; First posted 2018-05-08 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Uncertainty; Advanced Cancer; Family Members; Quality of Life
Keywords: uncertainty; caregivers; palliative care; nursing; Hospice and Palliative Care Nursing
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study proposes phase II in the development of randomized clinical trials for complex interventions, which refers to the development of an exploratory trial. This approach will be developed with participants randomly assigned to two groups (intervention and control) and pre-test and post-test measurements will be taken. The nursing intervention of this study is designed to be evaluated in terms of its viability, acceptability and preliminary effects in a health care institution with family caregivers of people with cancer in palliative care.
Who Masked: Participant
Masking Description: the participants in this study won't know if they are in the intervention group or in the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing intervention (Experimental): The experimental group will receive the Nursing intervention to reduce uncertainty in illness and increase quality of life in family caregivers of patients with cancer in palliative care
  Interventions: Other: Nursing intervention
- Conventional care (No Intervention): The control group will receive the nursing care conventionally given in the health care institution

INTERVENTIONS:
Other: Nursing intervention — The intervention was built on the components of the theory of uncertainty in illness and was designed to give in a face to face meeting with the caregiver education about advanced cancer in palliative care through an educational material.
  Educational material: The educational booklet has the purpose of giving information to the family caregiver about palliative care. This material aims to be an easily accessible resource to understand the palliative care of the cancer patient. In addition, this booklet will be used to ensure the standardization of the intervention during the face-to-face meeting with the participants and the investigator.
  Face-to-face meeting: The nursing intervention has a face-to-face meeting component between the investigator and the participant. This nursing educational session will be supported by the contents of the booklet and will have the purpose of discussing the contents of the booklet and resolving doubts on the part of the family caregivers.
  Arms: Nursing intervention

SUMMARY:
Background: The increase of chronic diseases has reached an increase in the suffering of advanced diseases and an inability of health care systems to give access to the population that suffers them. In this context are people with advanced cancer who are in palliative care and the family caregivers. Uncertainty in illness in palliative care and quality of life are two concepts that are altered in the patient's family caregiver in palliative care. Objective: to examine the feasibility and acceptability of a nursing intervention to reduce the uncertainty in illness and improve the quality of life of family caregivers of patients with cancer in palliative care. Methodology: Phase II clinical trial, the ratio of recruitment, follow-up of participants as well as satisfaction with the intervention will be evaluated as primary outcomes. As secondary outcomes, the possible effect of the intervention on the uncertainty in illness and the quality of life of the family caregiver will be evaluated. This study will be carry out in a health care institution in Medellin-Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Being the person responsible for the care of the person in palliative care most of the time
* Being over 18 years of age;
* Caring for a person who has a diagnosis of cancer stage IV, who is receiving palliative treatment for the disease and has an expectation longer than one month of life (determined by the physician)
* Being able to communicate in Spanish.

Exclusion Criteria:

* Being included in another institutional study of an educational nature
* Not knowing how to read
* Caring for another person with cancer before
* Have a significant cognitive disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | This variable will be measured during the process of recruitment of participants in the study that will be during a period of six months.
  this variable is defined as the proportion of eligible participants who agree to participate in the study, within the total of eligible participants. This variable will be measured with the Participant Recruitment Format.
Follow-up | this variable will be measured with the participants who complete the study, it will be measured with the participants after the intervention has finished within the framework of the study that will be six months.
  This variable is defined as the proportion of participants who entered the study and remained in the study until the post-intervention measurement within the total number of participants in the study. This variable will be measured with the Participation and Follow-up Format of the Participant.
Acceptability | this variable will be measured with the participants who complete the study in the intervention group. It will be measured after the intervention within the intervention group in the frame of execution of the study that will be six months.
  Refers to the perception that participants have of the intervention to address the problem presented in terms of being reasonable, adequate and convenient for its application in daily life and to meet their expectations. This variable will be measured with the Participant Satisfaction Questionnaire.

SECONDARY OUTCOMES:
Uncertainty in illness | this variable will be measure before and after the intervention. The time frame of this measurement will be first at day 1 before the intervention and 5 to 7 days after the intervention
  It is a cognitive state that is created when the individual can not adequately structure or categorize an event related to the disease due to insufficient signals to do so.
  the investigators will use the MISHEL UNCERTAINTY IN ILLNESS SCALE - FAMILY MEMBER FORM develop by Merle Mishel RN, PhD. This scale has 31 items with response options from 1 to 5, ranging from strongly disagree to strongly agree. This instrument in its original version has a structure of two factors. The first, Ambiguity with 19 items. The second, Complexity with 12. For populations with cancer the scale reports an alpha coefficient of between 0.77 to 0.91. The scale has a score of 31 to 150 points where the higher the score, the higher the level of uncertainty. The scale has evidence of transcultural adaptation and validity for the Colombian context.
Quality of life | this variable will be measure before and after the intervention. The time frame of this measurement will be first at day 1 before the intervention and 5 to 7 days after the intervention
  it is understood as the subjective perception that each subject has regarding their well-being. The scale measures the quality of life of the family caregiver of the person with cancer. In its original version it has a test-retest consistency of r = .89 and an internal consistency with an alpha value of 0.69. The scale has four dimensions, physical, psychological, social, spiritual well-being. The scale has a total of 37 items that are scored on a scale of 0 to 10, being 0 the worst result and 10 the best result. In its Spanish version it has a test-retest reliability of 0.88 and an internal consistency of 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia P Carreño, RN, MSc, PhD, Study Director — Universidad Nacional de Colombia

IPD SHARING:
Plan to Share IPD: Undecided
This item will be defined after the participants agree to share this information with other researchers. Even so if the information is blinded in terms of personal information for other investigations

REFERENCES:
- [Background] Northouse L, Kershaw T, Mood D, Schafenacker A. Effects of a family intervention on the quality of life of women with recurrent breast cancer and their family caregivers. Psychooncology. 2005 Jun;14(6):478-91. doi: 10.1002/pon.871. PMID 15599947
- [Background] Moore G, Collins A, Brand C, Gold M, Lethborg C, Murphy M, Sundararajan V, Philip J. Palliative and supportive care needs of patients with high-grade glioma and their carers: a systematic review of qualitative literature. Patient Educ Couns. 2013 May;91(2):141-53. doi: 10.1016/j.pec.2012.11.002. Epub 2012 Dec 5. PMID 23218925
- [Background] Henson LA, Higginson IJ, Daveson BA, Ellis-Smith C, Koffman J, Morgan M, Gao W; BuildCARE. 'I'll be in a safe place': a qualitative study of the decisions taken by people with advanced cancer to seek emergency department care. BMJ Open. 2016 Nov 2;6(11):e012134. doi: 10.1136/bmjopen-2016-012134. PMID 27807085
- [Background] Sparla A, Flach-Vorgang S, Villalobos M, Krug K, Kamradt M, Coulibaly K, Szecsenyi J, Thomas M, Gusset-Bahrer S, Ose D. Individual difficulties and resources - a qualitative analysis in patients with advanced lung cancer and their relatives. Patient Prefer Adherence. 2016 Oct 3;10:2021-2029. doi: 10.2147/PPA.S110667. eCollection 2016. PMID 27757022
- [Background] Chiou CP, Chung YC. Effectiveness of multimedia interactive patient education on knowledge, uncertainty and decision-making in patients with end-stage renal disease. J Clin Nurs. 2012 May;21(9-10):1223-31. doi: 10.1111/j.1365-2702.2011.03793.x. Epub 2011 Aug 26. PMID 21883569
- [Background] Scott AM, Martin SC, Stone AM, Brashers DE. Managing multiple goals in supportive interactions: using a normative theoretical approach to explain social support as uncertainty management for organ transplant patients. Health Commun. 2011 Jul-Aug;26(5):393-403. doi: 10.1080/10410236.2011.552479. Epub 2011 Jun 29. PMID 21409670
- [Background] Borneman T, Sun V, Williams AC, Fujinami R, Del Ferraro C, Burhenn PS, Irish T, Zachariah F, van Zyl C, Buga S. Support for Patients and Family Caregivers in Lung Cancer: Educational Components of an Interdisciplinary Palliative Care Intervention. J Hosp Palliat Nurs. 2015 Aug;17(4):309-318. doi: 10.1097/NJH.0000000000000165. PMID 26640416
- [Background] Bristowe K, Carey I, Hopper A, Shouls S, Prentice W, Caulkin R, Higginson IJ, Koffman J. Patient and carer experiences of clinical uncertainty and deterioration, in the face of limited reversibility: A comparative observational study of the AMBER care bundle. Palliat Med. 2015 Oct;29(9):797-807. doi: 10.1177/0269216315578990. Epub 2015 Mar 31. PMID 25829443